CLINICAL TRIAL: NCT06083064
Title: Protocol Based Selective Imaging Versus Routine Computed Tomography or Ultrasound in Suspected Appendicitis (PROSECCO)
Brief Title: Protocol Based Selective Imaging Versus Routine Computed Tomography or Ultrasound in Suspected Appendicitis
Acronym: PROSECCO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Panu Mentula, M.D., Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HUS/74/2023
Record Dates: First submitted 2023-10-05; First posted 2023-10-13 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Appendicitis
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Intervention Model Description: 1:1:1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Routine imaging (Active Comparator): Patients will have first abdominal ultrasound, and if findings are negative or inconclusive for appendicitis abdominal CT scan is made. If ultrasound is not available, CT scan can be the first imaging study. If appendicitis is found in the imaging study patient is scheduled for urgent laparoscopic appendectomy. Other patients are discharged or treated according to possible alternative diagnosis.
  Interventions: Diagnostic Test: Abdominal imaging
- Adult Appendicitis Score based selective imaging (Experimental): Adult Appendicitis Score (AAS) is calculated as soon as possible. Patients with AAS 16 or higher are scheduled for urgent laparoscopic appendectomy. Patients with AAS 11- 15 will have abdominal imaging as in the group 1. If appendicitis is found in the imaging study patient is scheduled for urgent laparoscopic appendectomy. Patients with AAS 10 or less are discharged without imaging studies.
  Interventions: Other: Score based selective abdominal imaging
- Appendicitis Severity Score based observation with selective imaging using Adult Appendicitis Score (Experimental): Patients with Adult Appendicitis Score (AAS) 10 or less are discharged without imaging studies. Patients with AAS 11 or more are managed based on Appendicitis Severity Score (ASS). ASS is used to identify patients with low risk of complicated disease. Patients with high ASS (>4) are managed as patients in arm 2. Patients with low ASS (<=4) begin observation protocol where patients can leave hospital and they are re-evaluated with repeated scoring after 12-24 hours from randomization. After re-scoring patients may be discharged if AAS is below 16 and decreasing and ASS is below 5 or if AAS is below 11. If AAS is 16 or higher or increasing, patients are scheduled for urgent laparoscopic appendectomy. After observation period, patients with decreasing AAS between 11-15 and ASS higher than 4 or patients with stable AAS between 11-15 are send for imaging study.
  Interventions: Other: Score based selective observation combined with selective abdominal imaging

INTERVENTIONS:
Diagnostic Test: Abdominal imaging — Abdominal ultrasound and/or abdominal CT
  Arms: Routine imaging
Other: Score based selective abdominal imaging — Abdominal imaging is done selectively based on Adult Appendicitis Score
  Arms: Adult Appendicitis Score based selective imaging
Other: Score based selective observation combined with selective abdominal imaging — Observation based on Appendicitis Severity Score combined Adult Appendicitis Score based selective abdominal imaging
  Arms: Appendicitis Severity Score based observation with selective imaging using Adult Appendicitis Score

SUMMARY:
The goal of this clinical trial is to compare protocol based selective imaging to routine imaging in adult patients with suspected appendicitis. The main question[s] it aims to answer are:

* Does protocol based selective imaging using clinical scoring affect clinical outcome?
* Does protocol based selective observation combined with score based selective imaging affect clinical outcome?

Participants will be randomized into three groups:

* Selective imaging based on Adult Appendicitis Score
* Selective observation based on Appendicitis Severity Score combined with selective imaging based on Adult Appendicitis Score
* Routine imaging using ultrasound and/or computed tomography

Researchers will compare selective imaging groups separately with routine imaging to see if number of negative appendectomies or number of complicated appendicitis is not significantly increased.

ELIGIBILITY:
Inclusion Criteria:

- Suspicion of appendicitis

Exclusion Criteria:

* Time from symptom onset over 72 hours
* Age <18 years
* Pregnancy, ruled out by serum or urine HCG measurement in 18- to 49-year-old women
* CT-scan or ultrasound already done within the last 3 days (72 hours)
* Clinical suspicion of other disease or other reason to perform imaging study
* Recruited earlier to the same trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Negative appendectomy | Within 30 days from randomization
  Number of negative appendectomies (surgical removal of non-inflamed appendix)
Complicated appendicitis | Within 30 days from randomization
  Number of patients with complicated appendicitis (AAST grade 3 or higher)

SECONDARY OUTCOMES:
histologically proven appendicitis | Within 30 days from randomization
  Number of patients with histologically proven appendicitis undergoing surgery
CT scan | Within 30 days from randomization
  Number of patients having abdominal computed tomography
Adverse events | Within one year from randomization
  Number patients with of adverse events (surgical complications, surgical site infections or delayed significant diagnosis)
Appendicitis | Within 2 years from randomization
  Number of patients diagnosed with appendicitis
Quality of life (EQ-5D-5L index value) | During the first 30 days from randomization
  Quality of life determined by weekly EQ-5D-5L index values.
Quality of life (EQ-5D-5L EQ-VAS score) | During the first 30 days from randomization
  Quality of life determined by weekly EQ-5D-5L EQ-VAS score.
Costs in Euros | During the first 30 days from randomization
  Overall costs of diagnostics and treatment

CONTACTS AND LOCATIONS:
Overall Officials: Panu Mentula, MD, Principal Investigator — Helsinki University Central Hospital
Locations (3):
- Finland (3):
  - HUS, Jorvi Hospital, Espoo
  - HUS, Meilahti Hospital, Helsinki
  - HUS, Hyvinkää Hospital, Hyvinkää

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sammalkorpi HE, Mentula P, Leppaniemi A. A new adult appendicitis score improves diagnostic accuracy of acute appendicitis--a prospective study. BMC Gastroenterol. 2014 Jun 26;14:114. doi: 10.1186/1471-230X-14-114. PMID 24970111
- [Background] Lastunen KS, Leppaniemi AK, Mentula PJ. DIAgnostic iMaging or Observation in early equivocal appeNDicitis (DIAMOND): open-label, randomized clinical trial. Br J Surg. 2022 Jun 14;109(7):588-594. doi: 10.1093/bjs/znac120. PMID 35482016
- [Background] Atema JJ, van Rossem CC, Leeuwenburgh MM, Stoker J, Boermeester MA. Scoring system to distinguish uncomplicated from complicated acute appendicitis. Br J Surg. 2015 Jul;102(8):979-90. doi: 10.1002/bjs.9835. Epub 2015 May 12. PMID 25963411